CLINICAL TRIAL: NCT03906019
Title: Defining the Indications and Levels of Erector Spinae Plane Block in Pediatric Patients: A Retrospective Study About Our Current Experience
Brief Title: Indications of Erector Spinae Plane Block in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, Assistant Professor, Kocaeli University
Other Study IDs: GOKAEK 2019/85
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Pain
Keywords: erector spinae plane block; postoperative pain; pediatric patients
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ESP Block — Erector spinae plane block performed with 0,25% bupivacaine (0,5 mL/kg-max 20mL), under general anesthesia before the start of the surgery.
Diagnostic Test: FLACC score — For up to 7 years old patients, Face, Legs, Activity, Cry and Consolability (FLACC) scores during postoperative 24h period.
Diagnostic Test: NRS score — Patients older than 7 years, NRS scores during postoperative 24h period.

SUMMARY:
Patients who were operated by Department of Pediatric Surgery between the 1 September 2017 and 28 February 2019 and who received erector spinae plane blocks as a part of postoperative analgesia management will be scanned.

DETAILED DESCRIPTION:
There are a few randomized prospective studies of ESPB for its clinical effectiveness and all of them are in adults, except one. Also pediatric case reports are limited when compared to adults. We have been applying ESPB to our patients almost since from its first definition. But ESPB applications for pediatric patients, in our clinic, have started after a learning curve. Patients who were operated by Department of Pediatric Surgery between the 1 September 2017 and 28 February 2019 and who received erector spinae plane blocks as a part of postoperative analgesia management will be scanned.

Demographical data of the patient, patient position for the block, indication/surgery type, level of ESPB, unilateral or bilateral application, total volume applied, additional analgesic use, type of the analgesic if used will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were operated by Department of Pediatric Surgery

Exclusion Criteria:

* Incomplete patient forms

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients who were operated by Department of Pediatric Surgery between the 1 September 2017 and 28 February 2019 and who received erector spinae plane blocks as a part of postoperative analgesia management.
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale | preoperative 24th hour
  A NRS involves asking the patient to rate his or her pain from 0 to 10 (11 point scale) with the understanding that 0 is equal to no pain and 10 is equal to worst possible pain.
Face, Legs, Activity, Cry and Consolability Score | postoperative 24th hour
  The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

CONTACTS AND LOCATIONS:
Overall Officials: Can Aksu, Assistant Professor, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University Hospital, İzmit, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No